CLINICAL TRIAL: NCT04875065
Title: Healthy Aging Research Program (HARP): Engage Coaching Project for Latinos
Brief Title: Engage Coaching for Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Caroline Silva, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006126; P30AG064103 (NIH)
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Social Isolation; Loneliness; Caregiver Burnout
MeSH Terms: conditions — Social Isolation; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Engage Coaching (Experimental): Engage Coaching helps caregivers bolster motivation for increasing connectedness, teaches problem solving skills, and provides behavioral practice with social engagement. Up to 8 brief sessions (typically 30 minutes) are provided weekly over no more than three months.
  Interventions: Behavioral: Engage coaching

INTERVENTIONS:
Behavioral: Engage coaching — Participants will complete up to 8 weekly individual Social Engage psychotherapy sessions. Participants will be allotted up to 3 months to complete all sessions, a time-frame that allows for two weeks without meeting to address life stressors such as illnesses that may pop up. All sessions are provided via phone or videocall (Zoom). The first and last session are longer - up to 60 minutes if needed. Middle sessions are shorter (20-45 minutes). Engage is a stepped care psychotherapy in that the simplest strategy is taught first-action planning (a derivative of problem solving therapy)-and "barrier strategies" are added only if needed. Action plans are designed to address loneliness and social isolation in the context of caregiving demands.

SUMMARY:
This study asks: "what behavioral strategies are needed to help socially disconnected Hispanic/Latino caregivers with significant barriers to increasing connectedness?" This study uses a mixed methods approach to adapt a brief behavioral intervention-Social Engage psychotherapy-for use with socially disconnected Hispanic/Latino caregivers. This study is a single-arm clinical trial of Social Engage psychotherapy. We propose to enroll 10 participants for up to 8 weekly individual Social Engage psychotherapy sessions, over up to 3 months. Subjects will be aged 40 and older, and be caregivers for a community-dwelling family member with ADRD, living with (or in close proximity to) the family member with dementia, experiencing elevated caregiving distress and social disconnectedness.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 yrs;
2. Hispanic/Latino
3. English or Spanish speaking;
4. Caregiver for a community-dwelling family member with ADRD, living with (or in close proximity to) family member with dementia;
5. Endorse elevated caregiving distress as measured by a score of ≥ 11 on the 10-item Perceived Stress Scale (PSS-10) and/or a score of 5 or greater on the Modified Caregiver Strain Index (MCSI);
6. Endorse clinically significant loneliness as measured by a score of ≥ 6 on the UCLA Loneliness Scale: Short Form.
7. Has access to e-mail in order to complete the e-consent module in REDCap which will be used in this study.

Exclusion Criteria:

1. Primary language is not English or Spanish;
2. Recent or current psychosis;
3. Significant cognitive impairment on a cognitive screening measure at the HARP screening assessment;
4. Hearing problems that preclude completion of the intervention.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Quinones MM, Silva C, Ross C, Sorensen S, Serrano R, Van Orden K, Heffner K. Recruiting Socially Disconnected Latinos Caring for a Person with Alzheimer's Disease and Related Dementias During the COVID-19 Pandemic: Lessons Learned. Clin Gerontol. 2023 Apr 2:1-14. doi: 10.1080/07317115.2023.2197895. Online ahead of print. PMID 37005703
- [Result] Quinones-Cordero MM, Norton S, Rivas C, Gallagher-Thompson D, Silva C. Exploring the unmet needs of Latino dementia caregivers: a qualitative study. Gerontologist. 2025 Oct 22;65(11):gnaf191. doi: 10.1093/geront/gnaf191. PMID 40929145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engage Coaching
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Engage Coaching
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.554643 (11.207574)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Loneliness at Post Intervention
Description: The UCLA Loneliness Scale Version 3 will be used to assess self-reported loneliness. 20 items, rated as to how often the participant has felt a certain way in the prior month (e.g., "How often do you feel alone?") -- "never" (1), "rarely" (2), "sometimes" (3), or "often" (4). Higher scores indicate greater loneliness. However, some individual items must be reverse-coded so that higher total scores reflect greater loneliness (i.e., 1=4, 2=3, 3=2, 4=1). These items (e.g., "How often do you feel there are people you can turn to?") are items 1,5,6,9,10,15,16,19,20. Total scores range from 20 to 80, with higher scores representing a worse outcome (i.e., greater loneliness). Mean change in total scores (change = baseline intervention scores - post scores) will be reported.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage Coaching
Number analyzed (Participants) | 8
score on a scale
  Baseline | 51.125000 (10.273927)
  3 Month | 53.000000 (12.200703)
Statistical Analysis 1: Comparison: Engage Coaching; Test type: Superiority; Mean Difference (Net) = -1.875000, 95% CI 2-sided [-13.236780 to 9.486780], Standard Error of Mean 4.804899 — Higher scale scores indicate greater loneliness. Thus, Mean change in total score is calculated as change = baseline intervention scores - post score, so that positive change values indicate symptom improvement

2. Secondary Outcome: Change From Baseline in Social Functioning at Post Intervention
Description: Satisfaction with Social Roles and Activities (PROMIS) is a computerized adaptive test (CAT). It produces T scores with a mean of 50 and standard deviation of 10. Greater scores indicate better outcomes (i.e., greater satisfaction with social role and activities). Mean change in T scores (change = post intervention scores - baseline scores) will be reported.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Engage Coaching
Number analyzed (Participants) | 8
T-scores
  Baseline | 41.332143 (4.756507)
  3 Month | 41.875000 (8.179897)
Statistical Analysis 1: Comparison: Engage Coaching; Test type: Superiority; Median Difference (Final Values) = 0.542857, 95% CI 2-sided [-5.107769 to 6.193483], Standard Error of Mean 2.389651 — Higher scale scores indicate better social functioning. Thus, Mean change in total score is calculated as change = post intervention scores - baseline score, so that positive change values indicate symptom improvement

3. Secondary Outcome: Change From Baseline in Quality of Life: Social Relationships at Post Intervention
Description: The World Health Organization Quality-of-Life Scale: Brief Version (WHOQOL-BREF) is a 36-item measure of several domains (physical health, psychological health, social relationships, environment) of health related quality of life. Higher scores denote higher quality of life. Items are scored on a 1-5 Likert scale. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval for each domain. Mean change in Domain 3 (social relationships) scores (change = post intervention scores - baseline scores) will be reported.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engage Coaching
Number analyzed (Participants) | 8
units on a scale
  Baseline | 41.687500 (24.326554)
  3 Month | 42.250000 (21.332403)
Statistical Analysis 1: Comparison: Engage Coaching; Test type: Superiority; Mean Difference (Net) = 0.562500, 95% CI 2-sided [-11.678525 to 12.803525], Standard Error of Mean 5.176732 — Higher scale scores indicate better social relationship quality of life. Thus, Mean change in total score is calculated as change = post intervention scores - baseline score, so that positive change values indicate symptom improvement

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Engage Coaching
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT04875065/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT04875065/ICF_000.pdf